CLINICAL TRIAL: NCT04247828
Title: Adaptive and Individualized AAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altec Inc. (Industry)
Collaborators: Madonna Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAC Phase I
Record Dates: First submitted 2020-01-21; First posted 2020-01-30 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-02

CONDITIONS: Communication Disorders
Keywords: Communication; Severe Physical Impairments; Spinal Cord Injury
MeSH Terms: conditions — Communication Disorders; Communication; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental and Generic Communication Interfaces for AAC (Experimental): Receives both Experimental and Generic AAC systems to communicate. Each participant will receive both devices, with Experimental AAC presented first (Day 1) and Generic AAC presented second (Day 2; reference).
  Interventions: Device: Experimental AAC; Device: Generic AAC

INTERVENTIONS:
Device: Experimental AAC — Participant receives an AAC system comprising a single hybrid wearable sensor for head-mediated cursor control that is integrated with an adaptive and individualized keyboard to test communication performance.
Device: Generic AAC — Participant receives an AAC system comprising a single hybrid wearable sensor for head-mediated cursor control that is integrated with a generic QWERTY keyboard to test communication performance.

SUMMARY:
This project will test the feasibility of developing a smart augmentative or alternative communication (AAC) system that is effective in delivering communication capabilities that automatically adapt to the users' physical abilities.

DETAILED DESCRIPTION:
The diversity of the more than 1.3% of Americans who suffer from severe physical impairments (SPIs) preclude the use of common augmentative or alternative communication (AAC) solutions such as manual signs, gestures or interaction with a touchscreen for communication. This clinical trial will test the feasibility of developing a smart-AAC system designed using individually adaptive access methods and AAC interfaces to accommodate the unique manifestations of motor impairments specific to each user. The investigators will demonstrate the proof-of-concept that a single surface electromyographic (sEMG) and inertial measurement unit (IMU) hybrid sensor worn on the forehead can provide improvements in information transfer rate (ITR) and communication accuracy when integrated with an AAC interface that is optimized compared to a conventional (non-adaptable) interface for subjects with SPI.

ELIGIBILITY:
Inclusion Criteria:

Control Subjects:

* Adults and Children; >12yo
* Male or Female
* All participants will be: (a) able to spell, (b) able to follow 2-3 step directions, (c) have functional vision sufficient to read 40 point text
* No history of communication disorders;
* No history of neurological disorders affecting speech or head movement.

Subjects with SPI:

* Adults or Children; age>12yo
* Male or Female
* All participants will be: (a) able to spell, (b) able to follow 2-3 step directions, (c) have functional vision sufficient to read 40 point text, and (d) have a motor impairment that requires the use of an alternative access strategy to communicate and/or use technology.
* Current or prospective AAC user with complex communication needs representing a broad spectrum of developmental and acquired SPI disabilities resulting from high spinal cord injury, chronic Guillain-Barré syndrome, brain stem stroke, cerebral palsy, locked-in syndrome, among others;
* Sufficient head control and voluntary facial muscle activation (on the basis of clinical evaluation by Dr. Susan Fager and her team) to use the proposed wearable EMG/IMU sensor for the purposes of this study;
* Evidence of at least partial voluntary head movement in at least 2 degrees of freedom (Individual differences in providing controlled movements of the head in various degrees of freedom due to their disease or trauma is not only acceptable but desirable);
* Sufficient stamina and developmental maturity (on the basis of clinical evaluation by Dr. Susan Fager) to attend to the approximately 1-hour protocol outlined in Aims 1 and 3 without excess fatigue or distraction;
* Availability for at least 3-4 testing sessions over the study period;
* No medical or safety restrictions of active head and neck movement (as determined by Dr. Susan Fager in consultation with her clinical team);
* Clinical evidence of preserved cognition by a score of 0 or 1 on NIHSS Consciousness and Communication item;
* Ability to voluntarily blink eyes or raise eyebrows on command.

Exclusion Criteria:

Control Subjects

* Non-English speaker;
* Inability to follow simple instructions in English;
* Restricted ROM of the head or neck;
* Pain with head movement
* Medical history of cardiac or respiratory complications, or disorders that would place the subject at risk for conducting the different motor activities;
* Skin disorders that result in open lesions or hyper-sensitive/fragile skin on the forehead, preventing the use of medical-grade adhesive tapes to secure the sensors to the skin;
* Unable to provide informed consent in English.

Subjects with SPI

* Non-English speaker;
* Inability to follow simple instructions in English;
* Medical history of musculoskeletal conditions (arthritis, spondylosis, etc.) that severely limit head movement or causes pain on head movement;
* Restricted active or passive rotation of head and neck resulting from unstable vertebral, spinal cord, or nerve roots that places the subject at risk;
* Medical history of cardiac or respiratory complications, or similar disorders that would severely reduce stamina and/or place the subject at risk for conducting the different motor activities;
* Skin disorders that result in open lesions or hyper-sensitive/fragile skin on the forehead, preventing the use of medical-grade adhesive tapes to secure the sensors to the skin;
* Unable to provide informed consent in English.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Contessa, PhD, Principal Investigator — Altec Inc.
Locations (2):
- United States (2):
  - Altec Inc., Natick, Massachusetts
  - Madonna Rehabilitation Hospital Institute for Rehabilitation Science and Engineering, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be made available within 6 months of study completion.
Access Criteria: Data access request will be made through conferencing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between January 6, 2020 and August 26, 2021.
Period: Overall Study
Arm/Group | Experimental and Generic Communication Interfaces for AAC
Started | 30
Started - Controls | 19
Started - Participants With SPI | 11
Completed | 21 (16 controls and 5 participants with SPI completed the study)
Not Completed | 9
Not completed — covid-19 mandated patient recruitment restrictions | 9

BASELINE CHARACTERISTICS:
Arm/Group | Experimental and Generic Communication Interfaces for AAC
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Movement Time
Description: Time needed to navigate a cursor to and select a target on a computer screen by control of head movement and facial muscle contractions for each AAC device, wherein lower movement times equate to better performance.
Time Frame: 1 Day
Population: All participants (control, SPI) experienced both the Experimental AAC (Day 1) and Generic AAC (reference, Day 2) devices. Of N=30 participants, N=9 were not analyzed as they could not complete the study protocol due to COVID-19 mandated restrictions in participant recruitment.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Experimental and Generic Communication Interfaces for AAC
Number analyzed (Participants) | 21
Seconds
  Experimental AAC | 2.5 (1.9)
  Generic AAC | 2.9 (2.0)

2. Primary Outcome: Path-to-Target Movement Variability
Description: Path smoothness relative to the optimal, straight path between targets on a computer screen by control of head movement and facial muscle contractions for each AAC device. Variability is estimated as a distance of pixels as estimated from a computer screen operating with a resolution of 1920 pixels x 1080 pixels, wherein smaller variability scores equate to better performance.
Time Frame: 1 Day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Experimental and Generic Communication Interfaces for AAC
Number analyzed (Participants) | 21
pixels
  Experimental AAC | 49.7 (9.4)
  Generic AAC | 74.0 (9.5)

3. Primary Outcome: Target Selection Accuracy
Description: Percentage of accurate selections of targets on a computer screen by control of head movement and facial muscle contractions for each AAC device, wherein higher accuracy scores equate to better performance.
Time Frame: 1 Day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Accurate Target Selections
Arm/Group | Experimental and Generic Communication Interfaces for AAC
Number analyzed (Participants) | 21
Percentage of Accurate Target Selections
  Experimental AAC | 96.3 (6.3)
  Generic AAC | 94.5 (9.8)

4. Primary Outcome: Information Transfer Rate
Description: Human motor performance relative to the speed and accuracy of cursor-to-target movements on a computer screen by control of head movement and facial muscle contractions for each AAC device, wherein higher information transfer rates equate to better performance.
Time Frame: 1 Day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bits/min
Arm/Group | Experimental and Generic Communication Interfaces for AAC
Number analyzed (Participants) | 21
Bits/min
  Experimental AAC | 45.8 (20.0)
  Generic AAC | 36.6 (16.2)

5. Primary Outcome: AAC Device Usability
Description: Self-report of perceived AAC device usability as captured via a Likert scale anchored from 1 ("very difficult") to 7 ("very easy"), wherein higher usability scores equate to better performance.
Time Frame: 1 Day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental and Generic Communication Interfaces for AAC
Number analyzed (Participants) | 21
units on a scale
  Experimentanl AAC | 4.7 (1.7)
  Generic AAC | 4.3 (2.9)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Experimental and Generic Communication Interfaces for AAC
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Not all recruited patients could complete the study protocol due to mandated patient recruitment restrictions resulting from the covid-19 emergency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT04247828/Prot_SAP_000.pdf